CLINICAL TRIAL: NCT01290731
Title: A Phase III, Open-label Trial in Japan to Investigate the Efficacy and Safety of TMC435 as Part of a Treatment Regimen Including Peginterferon Alfa-2a and Ribavirin in Genotype 1, Hepatitis C-infected Subjects Who Relapsed After Previous IFN-based Therapy
Brief Title: A Study of TMC435 in Genotype 1, Hepatitis C-infected Patients Who Relapsed After Previous Interferon (IFN)-Based Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017698; TMC435HPC3008 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Hepatitis C virus; Interferon Alfa-2a; Ribavirin; Viral RNA
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC435 100 mg 12 Wks + PR24/48 (Experimental): Participants will receive TMC435 100 mg once daily with PegIFNα-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24 (PR 24). Treatment will be stopped at Week 24 in participants who achieve plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels less than (<) 1.2 log10 IU/mL detectable or undetectable of at Week 4, and undetectable HCV RNA levels at Week 12. All other participants will continue PR until Week 48 (PR 48).
  Interventions: Drug: TMC435; Drug: Pegylated interferon (pegIFN alpha-2a); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: TMC435 — 100-mg capsule once daily for 12 weeks
Drug: Pegylated interferon (pegIFN alpha-2a) — 180 mcg injected subcutaneously (by a syringe under the skin) once weekly for 12 to 36 weeks (or until Week 48).
  Other Names: PEGASYS
Drug: Ribavirin (RBV) — 200-mg tablets (daily dose: 600-1000 mg) taken orally (by mouth) two times a day for 12 to 36 weeks (or until Week 48).
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TMC435 in combination with peginterferon alfa-2a (PegIFNα-2a) and ribavirin in genotype 1 hepatitis C virus (HCV)-infected participants who relapsed after previous interferon (IFN)-based therapy in Japan.

DETAILED DESCRIPTION:
This is a single-arm study to evaluate the efficacy and safety of TMC435 in combination with the standard of care (SoC), PegIFNα-2a (P) and ribavirin (R), in adult, genotype 1 HCV-infected participants who relapsed after previous IFN-based therapy in Japan. The study objective is to evaluate the efficacy of TMC435 by the percentage of participants with undetectable HCV ribonucleic acid (RNA). Participants will receive 12 weeks of treatment with TMC435 (100 mg) once daily plus PR followed by 12 or 36 weeks of treatment with PR. TMC435 is a 100-mg capsule and will be taken orally (via the mouth). Treatment with PR will last 24 or 48 weeks. Pegylated interferon is supplied as a vial containing 1.0 mL solution with 180 µg PegIFNα-2a and will be injected by a syringe under the skin once weekly. Ribavirin is given as 200-mg tablets (daily dose: 600-1000 mg), taken orally two times a day after meals. The participants will receive oral capsules of TMC435 (100 mg) once daily up to Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have chronic genotype 1 HCV with HCV RNA level >= 5.0 log10 IU/mL
* Participant relapsed after previous IFN-based therapy
* Participant must be willing to use contraceptive measures from the time of informed consent to 6 months after last dose of study medication.

Exclusion Criteria:

* Co-infection with any other HCV genotype or co-infection with the human immunodeficiency virus (HIV)
* Diagnosed with hepatic cirrhosis or hepatic failure
* A medical condition which is a contraindication to pegIFN or ribavirin therapy
* History of, or any current medical condition, which could impact the safety of the patient in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (10):
- Japan (10):
  - Hiroshima
  - Ichikawa
  - Kagoshima
  - Matsumoto
  - Musashino
  - Ohmura
  - Osaka
  - Sapporo
  - Suita
  - Touon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 22-Dec-2010 to 13-Aug-2012 and recruited participants with chronic Hepatitis C Virus (HCV) infection from 12 study centers in Japan. A total of 49 participants with chronic genotype 1 HCV infection were randomized and started treatment. A total of 48 participants completed the study.
Pre-assignment Details: HCV-infected participants who received at least 24 weeks of interferon (IFN)-based therapy and relapsed within 1 year after the last medication intake received treatment with TMC435 100 mg once daily with PegIFN alpha-2a and ribavirin (PR) until Week 12,followed by PR until Week 24/48 based on response-guided treatment (RGT) guidelines.
Groups:
- TMC435 100 mg 12 Wks + PR 24/48: Participants received TMC435 100 mg once daily with PegIFNa-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24 (PR 24). Treatment was to be stopped at Week 24 in participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants continued PR until Week 48 (PR 48).
Period: Overall Study
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48
Started | 49
Completed | 48
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 61 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a Sustained Virologic Response 12 Weeks After the Actual End of Treatment (SVR12)
Description: The table below shows the percentage of participants with an SVR12 defined as participants with undetectable plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) at the end of treatment (Week 24 or 48) who also had undetectable plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) 12 weeks after the last dose of treatment (Week 36 or 60).
Time Frame: Week 36 or 60
Population: The Full Analysis Set (FAS) consisted of all participants who received at least one dose of study drug during the study except for those who did not meet the major eligibility criteria for the study and participants who did not have efficacy data available after treatment with study medication.
Measure: Number; unit: Percentage of participants
Groups:
- TMC435 100 mg 12 Wks + PR24/48: Participants received TMC435 100 mg once daily with PegIFNα-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24 (PR 24). Treatment was to be stopped at Week 24 in participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable of at Week 4, and undetectable HCV RNA levels at Week 12. All other participants continued PR until Week 48 (PR 48).
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
Percentage of participants | 95.9

2. Secondary Outcome: The Percentage of Participants With a Sustained Virologic Response 24 Weeks After the Actual End of Treatment (SVR24)
Description: The table below shows the percentage of participants with a SVR24 defined as participants with undetectable plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) at the end of treatment (Week 24 or 48) and at 24 weeks after the last dose of treatment (Week 48 or 72).
Time Frame: Week 48 or 60
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
Percentage of participants | 89.8

3. Secondary Outcome: The Percentage of Participants Who Achieved a Greater Than or Equal to 2 log10 IU/mL Drop From Baseline in Plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) at Each Time Point During Treatment and Follow-up
Description: The table below shows the percentage of participants with greater than or equal to 2 log10 IU/mL drop from baseline in plasma HCV RNA at each time point during treatment, at the end of treatment (Week 24 or 48), and post-treatment follow-up.
Time Frame: Days 3 and 7, Weeks 2, 3, 4, 8, 12, 16, 20, 24, 28, 36, 48, 60, 72, EOT, and follow-up (FU) Weeks 4, 12, and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
Percentage of participants
  Day 3 | 93.9
  Day 7 | 100.0
  Week 2 | 100.0
  Week 3 | 98.0
  Week 4 | 100.0
  Week 8 | 100.0
  Week 12 | 100.0
  Week 16 | 98.0
  Week 20 | 100.0
  Week 24 | 95.9
  Week 28 | 100.0
  Week 36 | 93.9
  Week 48 | 89.8
  Week 60 | 89.8
  Week 72 | 89.8
  EOT | 100
  FU Week 4 | 100
  FU Week 12 | 95.9
  FU Week 24 | 91.8

4. Secondary Outcome: The Percentage of Participants With Undetectable Plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) During Treatment and at the End of Treatment (EOT)
Description: The table below shows the percentage of participants with undetectable HCV RNA (defined as less than 1.2 log10 IU/mL during treatment at Weeks 4, 12, 24, 36, 48, 60, 72, and at EOT [Week 24 or 48]).
Time Frame: Weeks 4, 12, 24, 36, 48, 60, 72, and at EOT
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
Percentage of participants
  Week 4 | 81.6
  Week 12 | 100.0
  Week 24 | 95.9
  Week 36 | 91.8
  Week 48 | 89.8
  Week 60 | 89.8
  Week 72 | 89.8
  EOT | 100.0

5. Secondary Outcome: The Number of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as a confirmed increase of greater than 1 log10 IU/mL in plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels from the lowest level reached or a confirmed value of plasma HCV RNA of > 2.0 log10 IU/mL in particpants whose plasma HCV RNA level had previously been below 1.2 log10 IU/mL detectable or undetectable during the treatment period. The table below shows that no viral breakthrough was noted in any participants during the treatment period of the study.
Time Frame: Day 1 until end of treatment (EOT [Week 24 or 48])
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
Participants | 0

6. Secondary Outcome: The Number of Participants Demonstrating Viral Relapse
Description: The table below shows the number of participants who demonstrated viral relapse, defined as undetectable Hepatitis C Virus Ribonucleic Acid (HCV RNA) at end of treatment (EOT) and detectable HCV RNA during follow-up or detectable HCV RNA at the time points of sustained virologic response (SVR) assessment . The incidence of viral relapse was calculated for participants with undetectable HCV RNA levels at EOT and with at least one follow-up HCV RNA measurement.
Time Frame: Up to 72 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
Participants | 4

7. Secondary Outcome: Plasma Concentrations of TMC435
Description: The table below shows median (range) TMC435 predose plasma concentration (C0h) values and the TMC435 maximum plasma concentration (Cmax) values for all participants who received TMC435 for up to 12 weeks. "Overall" is the median exposure estimate using all available data for each participant in the study.Sparse blood samples were collected during the study (blood sampling times were 3 and 5 hours post- dose at Week 2 and Week 8 and pre-dose and 2 hours post-dose at Week 4 and Week 12).
Time Frame: Overall (blood sampling times were 3 and 5 hours post- dose at Week 2 and Week 8 and pre-dose and 2 hours post-dose at Week 4 and Week 12)
Population: Pharmacokinetic (PK) analysis was performed in the PK population defined as all participants from whom sparse blood samples were drawn and who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
ng/mL
  C0h | 1822 [145 to 10693]
  Cmax | 3440 [1545 to 12273]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hrs (AUC24h) for TMC435
Description: The table below shows the median (range) AUC24h values for TMC435 for all participants who received TMC435 for up to 12 weeks. "Overall" is the median exposure estimate using all available data for each participant in the study. Sparse blood samples were collected during the study (blood sampling times were 3 and 5 hours post- dose at Week 2 and Week 8 and pre-dose and 2 hours post-dose at Week 4 and Week 12).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: ng.h/mL
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 49
ng.h/mL | 63261 [16480 to 276230]

9. Secondary Outcome: The Number of Participants With Abnormal Alanine Aminotransferase (ALT) Levels at Baseline Who Achieved Normal ALT Levels at the End of Treatment (EOT)
Description: The table below shows the number of participants with abnormal ALT levels at baseline (Day 1) who achieved normalization of ALT levels (defined as an ALT value less than or equal to the Upper Limit of Normality [ie, 40 IU/mL] at EOT). At baseline, 15/49 participants had abnormal ALT levels.
Time Frame: EOT (Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48
Number analyzed (Participants) | 15
Participants | 11

ADVERSE EVENTS:
Time Frame: Up to approximately 28 weeks (includes all serious and other adverse events that newly occurred or worsened after treatment with TMC435, PegIFNα-2b or ribavirin, until the end date of the last study medication intake + 28 days)
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48
Serious Adverse Events (participants affected / at risk) | 6/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100 mg 12 Wks + PR 24/48 (N=49)
Appendicitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100 mg 12 Wks + PR 24/48 (N=49)
Pyrexia (General disorders) | 36
Malaise (General disorders) | 22
Injection site reaction (General disorders) | 11
Fatigue (General disorders) | 4
Neutrophil count decreased (Investigations) | 30
White blood cell count decreased (Investigations) | 30
Platelet count decreased (Investigations) | 22
Haemoglobin decreased (Investigations) | 20
Haematocrit decreased (Investigations) | 13
Red blood cell count decreased (Investigations) | 11
Blood triglycerides increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 7
Weight decreased (Investigations) | 7
Blood calcium decreased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 5
Blood albumin decreased (Investigations) | 4
Blood cholesterol decreased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 4
High density lipoprotein decreased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Lipase increased (Investigations) | 3
Monocyte percentage increased (Investigations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 19
Alopecia (Skin and subcutaneous tissue disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 16
Dry skin (Skin and subcutaneous tissue disorders) | 8
Eczema (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 25
Dysgeusia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 22
Leukopenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 4
Retinal exudates (Eye disorders) | 5
Retinal haemorrhage (Eye disorders) | 3
Nasopharyngitis (Infections and infestations) | 5
Insomnia (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.